CLINICAL TRIAL: NCT02301013
Title: Are Unsatisfying Results After TVT and TOT Operations Associated With Increased Urethral Mobility
Brief Title: Impact of Urethral Mobility on the Success of Sling Operations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Agahan Han,MD, MD, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM01
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urinary incontience surgery (Experimental): Patients who is between 25 to 70 years old and positive stress test and have TVT or TOT operations with diagnoses of stress urinary incontinence and mixed urinary incontinence .
  Interventions: Procedure: Urinary incontience surgery; Drug: 300 cc saline

INTERVENTIONS:
Procedure: Urinary incontience surgery — Surgery for stress or mixed urinary incontience
Drug: 300 cc saline

SUMMARY:
Main objective is to evaluate the relation between the increased urethral mobility and unsuccessful treatment after TVT and TOT operations.

140 patients will be included in the research who are planned to have TVT and TOT operations with SUI and MUI diagnoses.Female patients of 25 to 70 years of age who are positive for stress test will be included.

All patients will be questioned for parity, body mass index, menopausal state, medical history, and examined for POP-Q stage, urodynamy, stress test, UDI 6, IIQ7 and with transperineal sonography preoperatively. "Passive mobility angle" and "active mobility angle" will be measured.

The relationship between passive mobility angle or active mobility angle and success of sling operations will be determined in this study.

DETAILED DESCRIPTION:
Transperineal sonography will be performed in a 300 cc filled bladder state, on a horizon which connects the lower margin of the pubic bone and the lower side of the urethral part of the bladder. First measurement will be done on litotomy position in resting state, second on 45 degrees reverse trandelenburg position in resting state and third one on 45 degrees reverse trandelenburg position in maximal valsalva straining state. The alteration between the angles measured at resting litotomy position and the resting reverse trandelenburg position is named as "passive mobility angle" (trigger gap) and the angle measured between the trigger gap and maximal valsalva state is named as "active mobility angle". Furthermore, post voiding residues have also been measured by transperineal ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* 140 patients will be included in the research who are planned to have TVT and TOT operations with SUI and MUI diagnoses between March 1, 2013 and January 1, 2015 in Kanuni Sultan Suleyman Medical Research and Educational Hospital.

Exclusion Criteria:

* Patients with level 3 or higher level of uterine descensus, previous urinary incontinence surgery, overactive bladder and who are unwilling for randomization will not been included.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Subjective Success of Sling Operations | 6 months
  Patients whose postoperative UDI-6 and IIQ-7 scores lower than 10 will described as success of sling operations

SECONDARY OUTCOMES:
Objective Success of Sling Operations | 6 months
  A patient with a bladder filled 300 cc saline will cough and if no leakage of urine,the patient will be described as ''cured''.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)